CLINICAL TRIAL: NCT01827007
Title: Assessment of Fluid Responsiveness by Elevation of PEEP in Patients With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Erika Wilkman, M.D, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS469/E6/05
Record Dates: First submitted 2013-04-02; First posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Septic Shock
Keywords: norepinephrine infusion; under 48 hours in ICU
MeSH Terms: conditions — Shock, Septic | interventions — Polygeline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm, elevation of PEEP (Experimental)
  Interventions: Other: Volume expansion with gelofusine

INTERVENTIONS:
Other: Volume expansion with gelofusine

SUMMARY:
The aim of the study is to evaluate whether fluid responsiveness of the critically ill patient can be assessed by analysing the PEEP-induced hemodynamic effects to systolic blood pressure, pulse pressure, aortic blood flow, aortic time-velocity integral and left ventricular end diastolic area measured with transesophageal echocardiography (PEEP-test). The chances are compared to increase of CI after volume expansion (gold standard). In clinical practise, it would be especially relevant if PEEP-induced changes in arterial pressure variations could be used in evaluation of volume status and fluid responsiveness. However, as ECHO-derived variables are used in greater extent to guide the treatment with inappropriate evidence, the simultaneous registration of ECHO-derived hemodynamic measurements is essential in the study design.

ELIGIBILITY:
Inclusion Criteria:• Written informed consent by patient or relative

* Time in ICU < 48 hours
* Septic shock
* Pulmonary artery catheter and radial arterial catheter
* Age 18 - 75 years
* Sinus rhythm
* Need for norepinephrine over 0.1 ug/kg/min but otherwise hemodynamically stable i.e no need to change the dose over the last 15min period before the study
* Mechanical ventilation with sedation
* Pwcp <18 mmHg

Exclusion Criteria:

* Contraindication to elevation of PEEP ( elevated intracranial pressure, pulmonary hypertension or other contraindication )
* Contraindication to fluid challenge
* Contraindication to TEE
* Previous heart failure, heart valve stenosis of insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Hemodynamic changes indicating fluid responsiveness assessed during elevation of PEEP. Change in mean arterial pressure or aortic velocity time integral. | Measurement of hemodynamic variables at timepoints 0, 10,20, 60 minutes
  Measurement of hemodynamic variables using a pulmonary catheter and transesophageal echocardiography at baseline PEEP 10, during elevation of PEEP and after volume challenge at PEEP 10 cmH2O

SECONDARY OUTCOMES:
Pulmonary function and oxygenation | 0,10,20,60 minutes, at PEEP 10, 20,10 cmH2O and after fluid expansion PEEP10 cmH2O

OTHER OUTCOMES:
blood gas sample, for assessment of pH, base excess and blood lactate | 0, 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Erika Wilkman, M.D, Principal Investigator — Anesthesia and Intensive Care, Department of Surgery
Locations (1):
- Intensive Care Unit 20, Meilahti Hospital, Helsinki, HUS, Finland